CLINICAL TRIAL: NCT00217659
Title: A Phase II Study of Goserelin Plus Anastrozole for the Treatment of Male Patients With Hormone-Receptor Positive Metastatic or Recurrent Breast Cancer
Brief Title: S0511, Goserelin and Anastrozole in Treating Men With Recurrent or Metastatic Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: poor accrual
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000442919; S0511 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2013-01

CONDITIONS: Breast Cancer
Keywords: male breast cancer; recurrent breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Anastrozole; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: anastrozole
Drug: goserelin acetate

SUMMARY:
RATIONALE: Estrogen can cause the growth of breast cancer cells. Hormone therapy using goserelin and anastrozole may fight breast cancer by blocking the use of estrogen by the tumor cells. Giving goserelin together with anastrozole may be an effective treatment for male breast cancer.

PURPOSE: This phase II trial is studying how well giving goserelin together with anastrozole works in treating men with recurrent or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the progression-free survival (PFS) of men with estrogen receptor- or progesterone receptor-positive recurrent or metastatic breast cancer treated with goserelin and anastrozole.
* Determine the overall survival of patients treated with this regimen.
* Determine the overall objective tumor response rate (confirmed and unconfirmed, complete and partial) in patients with measurable disease treated with this regimen.
* Correlate prostate specific antigen (PSA), testosterone, estradiol, estrone, estrone sulfate, follicle-stimulating hormone, luteinizing hormone, and dehydroepiandrosterone levels with PFS and response in patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive goserelin subcutaneously on day 1 and oral anastrozole on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at approximately 4-6 weeks and then every 3-6 months for up to 3 years.

PROJECTED ACCRUAL: A total of 56 patients will be accrued for this study within 48 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed breast cancer

  * Recurrent or metastatic (stage IV) disease

    * Patients with a local regional recurrence, including axillary and/or chest wall involvement, are eligible
* Measurable or non-measurable disease
* Brain metastases allowed provided they have been treated with surgery or radiotherapy AND have remained stable for ≥ 3 months
* Hormone receptor status:

  * Estrogen receptor- OR progesterone receptor- positive disease by standard immunohistochemical techniques

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Male

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* No evidence of severe or uncontrolled hepatic disease

Renal

* No evidence of severe or uncontrolled renal disease

Cardiovascular

* No evidence of severe or uncontrolled cardiac disease

Pulmonary

* No evidence of severe or uncontrolled respiratory disease

Other

* Fertile patients must use effective barrier-method contraception during and for 12 weeks after the completion of study treatment
* No known HIV positivity
* Able to receive oral medication

  * Patients with a gastrointestinal tube are eligible
* No known hypersensitivity to luteinizing hormone-releasing hormone (LHRH), LHRH agonist analogues, or any components of the study drugs
* No active infection requiring systemic therapy
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer
* No evidence of other severe or uncontrolled systemic disease

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent prophylactic filgrastim (G-CSF) or other hematopoietic growth factors

Chemotherapy

* At least 14 days since prior chemotherapy for this cancer and recovered
* No more than 1 prior chemotherapy regimen for metastatic disease
* No concurrent chemotherapy

Endocrine therapy

* At least 14 days since prior hormonal therapy for this cancer and recovered
* Prior tamoxifen allowed
* No prior gonadotropin-releasing hormone antagonist, aromatase inhibitors, or fulvestrant
* No other concurrent hormonal therapy (e.g., estrogen-based therapies)

Radiotherapy

* See Disease Characteristics
* At least 14 days since prior radiotherapy for this cancer and recovered
* No concurrent radiotherapy

Surgery

* See Disease Characteristics

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-09; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS)
Overall survival
Overall objective tumor response rate (confirmed and unconfirmed, complete and partial)
Correlation of prostate specific antigen, testosterone, estradiol, estrone, estrone sulfate, follicle-stimulating hormone, luteinizing hormone, and dehydroepiandrosterone levels with PFS
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Zeina Nahleh, MD — Barrett Cancer Center; Abdul-Rahman Jazieh, MD, MPH — Barrett Cancer Center; Robert B. Livingston, MD — University of Washington; Gabriel N. Hortobagyi, MD, FACP — M.D. Anderson Cancer Center
Locations (57):
- United States (57):
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - Montrose Memorial Hospital Cancer Center, Montrose, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Community Oncology Group at Cleveland Clinic Cancer Center, Independence, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - AnMed Health Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming